CLINICAL TRIAL: NCT00236691
Title: Double-Blind, Parallel Comparison of Three Doses of Topiramate and Placebo in Refractory Partial Epilepsy
Brief Title: A Study of the Efficacy and Safety of Topiramate as add-on Therapy in the Treatment of Epilepsy Patients With Difficult to Treat, Partial-onset Seizures.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005452
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Epilepsy; Epilepsies, Partial; Seizures
Keywords: topiramate; epilepsy; partial epilepsies; partial epilepsy; seizures; epileptic seizures; partial seizure disorder; brain diseases
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Seizures; Brain Diseases | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of topiramate as add-on therapy in patients with difficult to control partial onset seizures who are taking one or two standard antiepileptic drugs.

DETAILED DESCRIPTION:
Epilepsy is characterized by seizures, which are abnormal electrical discharges in the brain that temporarily disrupt normal brain function. Seizures are classified as "generalized," originating in both sides of the brain simultaneously, or "partial-onset," starting in one area of the brain. Antiepilepsy medications, such as topiramate, are selected based on seizure type. This is a double-blind, placebo-controlled study to evaluate the efficacy and safety of topiramate as add-on therapy in patients with refractory partial epilepsy, that includes a baseline phase and a treatment phase in difficult to treat patients with partial epilepsy. During the baseline phase (12 weeks duration), patients receive one or two of the following standard antiepileptic drugs (AEDs): phenytoin, carbamazepine, phenobarbital, primidone, or valproic acid. Patients who continue to have seizures during treatment with standard AEDs proceed into the double-blind treatment phase. Patients then receive placebo or topiramate at a dosage of 100-milligrams (mg) twice daily, increasing to twice daily dosing at a maximum dose 600 mg/day, 800 mg/day, or 1000 mg/day, or maximum tolerated dose (depending on treatment group), through Week 18 (total duration of the double-blind phase), while continuing on their standard AED regimen. Assessments of effectiveness include the percent reduction in the average monthly seizure rate, percent of patients responding to treatment (having equal to or greater than 50% reduction in seizure rate), and the patient's and investigator's global assessments of medication at end of study. Safety assessments include the incidence of adverse events throughout the study, clinical laboratory tests (hematology, serum chemistry, urinalysis), neurologic examinations, and vital sign measurements (blood pressure, pulse, temperature) weekly during the treatment phase. The study hypothesis is that topiramate, taken as add-on therapy to treatment with AEDs, will significantly reduce seizure frequency, compared with placebo, in patients with refractory partial epilepsy. In addition, it is hypothesized that topiramate is well-tolerated. Topiramate, 100 mg oral tablets, or matching placebo. Dosage begins at 100-mg twice daily and increases gradually to twice daily dosing at a maximum dose of 600, 800, or 1000 mg/day, and continues through Week 18 (total duration).

ELIGIBILITY:
Inclusion Criteria:

* History of simple or complex partial epilepsy that has been documented or witnessed
* during a 12-week baseline phase, patient must have at least 12 partial seizures while maintaining therapeutic levels of anti-epileptic drugs (AEDs)
* and have no more than one seizure-free interval of up to 3 weeks and none longer than 3 weeks
* good physical health.

Exclusion Criteria:

* Females who are capable of having children
* patients with treatable causes of seizures (for example, infections)
* patients with a progressive disorder of the nervous system
* patients with history of status epilepticus (repeated or prolonged seizures) while on antiepileptic therapy
* history of serious disease of the heart, liver, kidneys, gastrointestinal, metabolic, or endocrine system
* history of alcohol or drug abuse within one year prior to study initiation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 1988-07; Study Completion 1990-12 (Actual)

PRIMARY OUTCOMES:
Percent reduction in the average monthly seizure rate from baseline to end of treatment

SECONDARY OUTCOMES:
Percent of patients responding to treatment (>= 50% reduction in seizure rate from baseline to end of treatment); patient's and investigator's global assessments at end of study; incidence of adverse events and safety are evaluated throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the effectiveness and safety of topiramate in the treatment of patients with epilepsy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=643&filename=CR005452_CSR.pdf